CLINICAL TRIAL: NCT05737108
Title: A Clinical Trial on the Efficacy of Bilberry-containing Capsules for Dry Eye Mitigation
Brief Title: Bilberry-containing Capsules for Dry Eye Mitigation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Collaborators: Glory Kingdom Corporation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 111-73
Record Dates: First submitted 2022-11-18; First posted 2023-02-21 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2023-05

CONDITIONS: Dry Eye
Keywords: bilberry; anthocyanin; dry eye; eye sore; eye strain
MeSH Terms: conditions — Dry Eye Syndromes; Asthenopia | interventions — Vaccinium myrtillus extract; Pharmaceutical Preparations

STUDY DESIGN:
Intervention Model Description: Intervention with oral intakes of either test samples or placebo for 30 days, followed by a 20-day period of washout, and then crossover for another 30 days of either test samples or placebo.
Who Masked: Participant, Care Provider
Masking Description: Only investigators and outcomes assessors have knowledge on whether the samples given are tests or placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A-test samples (Experimental): This group will be given test bilberry capsule for 30 days and then have a washout period for 20 days.
  Interventions: Dietary Supplement: Bilberry capsule product; Dietary Supplement: Placebo(starch)
- Group A-placebo (Placebo Comparator): This group will be given placebo for 30 days and then have a washout period for 20 days.
  Interventions: Dietary Supplement: Bilberry capsule product; Dietary Supplement: Placebo(starch)

INTERVENTIONS:
Dietary Supplement: Bilberry capsule product — A specific bilberry capsule product, containing bilberry dried extracts at 23.2 mg and bilberry powder at 3.2 mg will be given to participants for oral intake for 30 days. 30 days of Bilberry capsule product or placebo with crossover to the other.
Dietary Supplement: Placebo(starch) — 30 days of placebo or Bilberry capsule product with crossover to the other.

SUMMARY:
This study investigates whether the oral intake of a bilberry capsule product may relieve dry eye symptoms. Participants will be aged between 20 - 65 years of age, with confirmed diagnosis of dry eye status. The participants will be assessed for several parameters and asked to take 4 bilberry capsules per day for 30 days. The parameters will include ocular surface health, tear volume, tear quality, intraocular pressure, and tear compositions. After the 30 days are completed, the participants will be assessed again for the same parameters.

DETAILED DESCRIPTION:
This investigation is a randomized, double-blind study. Subjects with confirmed diagnosis of dry eye are randomly assigned to group A or group B, and asked to orally intake 4 capsules of either bilberry product or placebo per day.The group A will have bilberry product for 30 days, have a 20-day washout period, and then have placebo for another 30 days. The group B will have placebo for 30 days, have a 20-day washout period, and then have bilberry product for another 30 days. All participants will be assessed for parameters, including intraocular pressure, ocular surface health, tear film breakup time (TBUT), tear volume (Schirmer's test), tear composition (Na+, K+, Cl- ions), tear osmolarity, ocular surface impression cytology, and ocular surface disease index (OSDI). The assessments are conducted immediately before the first 30-day and immediately after the second 30-day oral intake period. The parameters are used to compare and evaluate whether the bilberry product can relieve dry eye symptoms.

ELIGIBILITY:
Inclusion Criteria:

* aged between 20 and 65 years
* with Schirmer's test results between 5 - 10 mm or Tear Film Break Up Time less than 10 seconds
* Ocular Surface Disease Index more than 25

Exclusion Criteria:

* evident ocular diseases such as cornea disease, cataract, vitreous degeneration, glaucoma, and retinopathy.
* diabetes
* hypertension
* or other chronic diseases or belong to vulnerable groups(pregnancy woman, prisoner, ethical minorities, economic or educationally disadvantaged subjects, disabled individuals such as those at terminal stage of tumorigenesis, blindness, terminal ill individuals)

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-08-24 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change From Baseline of Schirmer's Test Value at Day 31 | on baseline and day31
  To assess tear secretion volume. The amount of tears are measured in total millimeters after 5 minutes has elapsed. Lower measurement indicates presence of dry eye disease.
Change From Baseline of Tear Film Breakup Time at Day 31 | on baseline and day31
  Tear Break-Up Time is a measurement in seconds of tear film stability. The shorter the Tear Break-Up Time, the lower the tear film stability. Less than 10 seconds = dry eye disease; lower score indicates worse disease.
Change From Baseline of Ocular Surface Index at Day 31 | on baseline and day31
  To assess the health status with Fluorescein stain. Scale ranges from 0 to 3, where grade 0 = None, 3 = Severe

SECONDARY OUTCOMES:
Change From Baseline of Tear Contents at Day 31 | on baseline and day31
  Determination of changes in osmolality and ion content for test groups of sample or placebo.
Change From Baseline of Ocular Surface Impression Cytology at Day 31 | on baseline and day31
  To assess the status of conjunctival goblet cells and epithelium.
Change From Baseline of Ocular Surface Disease Index Score at Day 31 | on baseline and day31
  A questionnaire to assess the health status on ocular surface, with higher scores indicating greater disability.
Change From Baseline of Intraocular Pressure at Day 31 | on baseline and day31
  To determine the effects of intervention on intraocular pressure.

CONTACTS AND LOCATIONS:
Overall Officials: David Pei-Cheng Lin, PhD, Principal Investigator — Chung Shan Medical University
Locations (1):
- Jen-Ai Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Masmali AM, Purslow C, Murphy PJ. The tear ferning test: a simple clinical technique to evaluate the ocular tear film. Clin Exp Optom. 2014 Sep;97(5):399-406. doi: 10.1111/cxo.12160. PMID 25138744
- [Background] The definition and classification of dry eye disease: report of the Definition and Classification Subcommittee of the International Dry Eye WorkShop (2007). Ocul Surf. 2007 Apr;5(2):75-92. doi: 10.1016/s1542-0124(12)70081-2. PMID 17508116
- [Background] Fox RI, Chan R, Michelson JB, Belmont JB, Michelson PE. Beneficial effect of artificial tears made with autologous serum in patients with keratoconjunctivitis sicca. Arthritis Rheum. 1984 Apr;27(4):459-61. doi: 10.1002/art.1780270415. No abstract available. PMID 6712760
- [Background] Wilson WS, Duncan AJ, Jay JL. Effect of benzalkonium chloride on the stability of the precorneal tear film in rabbit and man. Br J Ophthalmol. 1975 Nov;59(11):667-9. doi: 10.1136/bjo.59.11.667. PMID 1203224
- [Background] Brito-Zeron P, Ramos-Casals M; EULAR-SS task force group. Advances in the understanding and treatment of systemic complications in Sjogren's syndrome. Curr Opin Rheumatol. 2014 Sep;26(5):520-7. doi: 10.1097/BOR.0000000000000096. PMID 25050925
- [Background] Sullivan DA, Krenzer KL, Sullivan BD, Tolls DB, Toda I, Dana MR. Does androgen insufficiency cause lacrimal gland inflammation and aqueous tear deficiency? Invest Ophthalmol Vis Sci. 1999 May;40(6):1261-5. PMID 10235562
- [Background] Schrader S, Mircheff AK, Geerling G. Animal models of dry eye. Dev Ophthalmol. 2008;41:298-312. doi: 10.1159/000131097. PMID 18453777
- [Background] Ozawa Y, Kawashima M, Inoue S, Inagaki E, Suzuki A, Ooe E, Kobayashi S, Tsubota K. Bilberry extract supplementation for preventing eye fatigue in video display terminal workers. J Nutr Health Aging. 2015 May;19(5):548-54. doi: 10.1007/s12603-014-0573-6. PMID 25923485
- [Background] Kosehira M, Machida N, Kitaichi N. A 12-Week-Long Intake of Bilberry Extract (Vaccinium myrtillus L.) Improved Objective Findings of Ciliary Muscle Contraction of the Eye: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Comparison Trial. Nutrients. 2020 Feb 25;12(3):600. doi: 10.3390/nu12030600. PMID 32106548